CLINICAL TRIAL: NCT05930132
Title: The Role of Using the Submucosal Conchoplasty Technique for the Management of Concha Bullosa in Decreasing the Postoperative Middle Meatus Synechia Formation After Endoscopic Sinus Surgery: A Randomized Controlled Trial
Brief Title: The Role of the Submucosal Conchoplasty Technique in Improving the Postoperative Middle Meatus Outcome After ESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Waheed Elgendy, lecturer of otolaryngology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKSU50-9-22
Record Dates: First submitted 2023-06-14; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Endoscopic Sinus Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic lateral lamellectomy (Other): Regarding the lateral lamellectomy technique, the concha was locally infiltrated with adrenaline with a concentration of 1:200,000; the sickle knife was used to open the concha then the scissor was used to remove the lateral lamella with its covering mucosa in one block.
  No middle meatus packing was applied. Systemic antibiotics and steroids (0.5 mg / kg prednisolone) were given for two weeks after the surgery. The patients were instructed to use local nasal irrigations (2 ml of budesonide 0.5 mg / ml mixed with 250 ml of normal saline) two times daily for a month postoperatively. Patients were followed up at the end of each month throughout the six months follow-up period.
  Interventions: Procedure: classic lateral lamellectomy
- submucosal conchoplasty (Other): Regarding the submucosal conchoplasty technique, the concha was locally infiltrated with adrenaline with a concentration of 1:200,000. The mucosa was incised by blade 15 starting from the axilla posteriorly up to the attachment with the basal lamella. The mucosa covering the lateral lamella was dissected using the freer dissector. The lateral lamella was removed using a through cut forceps then the mucosa was repositioned. The bony skeleton of the medial lamella was preserved
  Interventions: Procedure: submucosal conchoplasty

INTERVENTIONS:
Procedure: submucosal conchoplasty — Regarding the submucosal conchoplasty technique, the concha was locally infiltrated with adrenaline with a concentration of 1:200,000. The mucosa was incised by blade 15 starting from the axilla posteriorly up to the attachment with the basal lamella. The mucosa covering the lateral lamella was dissected using the freer dissector. The lateral lamella was removed using a through cut forceps then the mucosa was repositioned. The bony skeleton of the medial lamella was preserved
  Arms: submucosal conchoplasty
Procedure: classic lateral lamellectomy — Regarding the lateral lamellectomy technique, the concha was locally infiltrated with adrenaline with a concentration of 1:200,000; the sickle knife was used to open the concha then the scissor was used to remove the lateral lamella with its covering mucosa in one block.
  No middle meatus packing was applied. Systemic antibiotics and steroids (0.5 mg / kg prednisolone) were given for two weeks after the surgery. The patients were instructed to use local nasal irrigations (2 ml of budesonide 0.5 mg / ml mixed with 250 ml of normal saline) two times daily for a month postoperatively. Patients were followed up at the end of each month throughout the six months follow-up period.
  Arms: classic lateral lamellectomy

SUMMARY:
The study aimed to compare the applicability of the classic lateral lamellectomy versus the submucosal conchoplasty techniques in managing the concha bullosa during and after ESS.

DETAILED DESCRIPTION:
The study included fifty-six patients with bilateral concha bullosa who were undergoing primary ESS for refractory chronic sinusitis. They were divided into two equal groups randomly. One group had the submucosal conchoplasty technique, and the other group had the lateral lamellectomy technique. The study compared the intraoperative findings including the time required for each technique and the amount of intraoperative bleeding. Furthermore, it compared the postoperative endoscopic outcome of the middle meatus and middle turbinate stability using the LKES and the POSE score. Also, the postoperative olfaction outcome was assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years
* patients diagnosed with chronic sinusitis based on the 2012 European Position Paper on Rhino-sinusitis and Nasal Polyps's criteria (EPOS 2012)
* patients presented by bilateral concha bullosa

Exclusion Criteria:

* patients below 18 years
* smokers
* patients with nasal polyps
* patients with primary ciliary dyskinesia
* patients with nasal masses
* revision cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
the clinical symptoms before and after the surgery through the Sino-nasal outcome test 22. (SNOT 22) | Patients were followed up at the end of six month after surgery ( change from baseline )
  The study assessed the clinical symptoms before and after the surgery through the Sino-nasal outcome test 22. (SNOT 22)

SECONDARY OUTCOMES:
the time of the technique | during the operation
  in minutes
the amount of bleeding | during the operation
  in cubic centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh university, Sakhā, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No